CLINICAL TRIAL: NCT07151534
Title: Investigation of the Relationship Between Body Awareness, Trunk Stabilization, and Upper Extremity Functionality in Individuals With Multiple Sclerosis
Brief Title: Body Awareness, Trunk Stability, and Arm Function in MS
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, Principal Investigator, Hacettepe University
Other Study IDs: Body Awareness
Record Dates: First submitted 2025-08-06; First posted 2025-09-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: body awareness; upper extremity; trunk stabilization; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis: Diagnosed with Multiple Sclerosis (MS) by a neurologist according to the McDonald criteria, aged 18 years or older, Expanded Disability Status Scale (EDSS) score of ≤ 5, Mini-Mental State Examination score of 24 or higher will be included in the study.
- Healthy: A control group consisting of healthy individuals matched with MS patients by age and sex will be included in the study.

SUMMARY:
The aim of this study is to investigate the relationship between body awareness, trunk stabilization, and upper extremity functionality in patients with Multiple Sclerosis (MS).

Hypotheses of the study:

H1: There is a significant relationship between body awareness and upper extremity functionality in patients with MS.

H2: There is a significant relationship between body awareness and trunk stabilization in patients with MS.

H3: Body awareness is reduced in patients with MS compared to healthy individuals.

H4: Trunk stabilization is reduced in patients with MS compared to healthy individuals.

H5: Upper extremity functionality is reduced in patients with MS compared to healthy individuals.

DETAILED DESCRIPTION:
Patients' demographic and disease-specific information will be recorded. Subsequently, body awareness, upper extremity functionality, and trunk stabilization will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Multiple Sclerosis (MS) by a neurologist according to the McDonald criteria
* Aged 18 years or older
* Expanded Disability Status Scale (EDSS) score ≤ 5
* Mini-Mental State Examination (MMSE) score ≥ 24

  * A control group consisting of healthy individuals matched with MS patients in terms of age and sex

Exclusion Criteria:

* Having a neurological disorder other than MS
* Having experienced a relapse and/or used corticosteroids in the past 3 months
* Having an orthopedic/systemic condition affecting the upper extremities or trunk
* Being pregnant
* Refusing to participate or not providing written informed consent

  * Healthy individuals who have an orthopedic/systemic condition affecting the upper extremities or trunk, who are pregnant, or who do not agree to participate and provide written informed consent will be excluded.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MS patients and healthy subjects with inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Body Awareness Questionnaire | up to 6 months
  To assess body awareness, the Body Awareness Questionnaire will be used.This questionnaire consists of 18 items, each scored on a scale from 1 to 7, and evaluates body awareness. Higher scores indicate better body awareness. The Turkish version has been validated and found to be reliable.
Body Awareness Rating Questionnaire | up to 6 months
  To assess body awareness,the Body Awareness Rating Questionnaire will be used. Body Awareness Rating Questionnaire:This questionnaire includes 24 items across 4 domains: function, mood, feeling/sensation, and awareness. Higher scores indicate better body awareness. The Turkish version has been validated and shown to be reliable.
Upper Extremity Functionality-Grip strength | up to 6 months
  Grip strength will be measured with a Jamar dynamometer. It will be performed three times bilaterally, and average values (kg) will be recorded.
Upper Extremity Functionality-Pinch strength | up to 6 months
  Pinch strengths will be assessed using a Baseline pinch gauge. It will be performed three times bilaterally, and average values (kg) will be recorded.
Upper Extremity Functionality-Nine Hole Peg Test (9HPT) | up to 6 months
  The 9HPT will evaluate hand dexterity by timing how quickly participants place and remove nine pegs. Each hand will be tested three times. It will be recorded in seconds. An average time ≥33.3 seconds will indicate dysfunction in MS patients.
Trunk Stabilization- Trunk Impairment Scale (TIS), | up to 6 months
  Trunk stabilization will be evaluated using the TIS.TIS: Assesses static/dynamic balance and trunk coordination (17 items, 0-23 points).
Trunk Stabilization-plank endurance test | up to 6 months
  Trunk stabilization will be evaluated using the plank endurance test. The test measures core endurance. Plank test: Time held in forearm plank recorded. It will be recorded in seconds.
Trunk Stabilization-side bridge test | up to 6 months
  Trunk stabilization will be evaluated using the side bridge test. The test measures core endurance Time held in side plank on both sides recorded.It will be recorded in seconds.
Trunk Stabilization-Modified Biering-Sorensen | up to 6 months
  Trunk stabilization will be evaluated using the Modified Biering-Sorensen test. The test measures core endurance. Time holding trunk in horizontal position prone over table edge. It will be recorded in seconds.
Trunk Stabilization-Trunk flexor test | up to 6 months
  Trunk stabilization will be evaluated using the Trunk flexor test test.The test measures core endurance. Time maintaining 60° trunk flexion with knees/hips at 90°. It will be recorded in seconds.
Trunk Stabilization-Sit up test | up to 6 months
  The 30-second Sit-up Test measures core strength. The person lies on their back with knees bent and feet on the floor. They do as many sit-ups as possible in 30 seconds, keeping proper form. The score is the number of correct sit-ups completed.
Trunk Stabilization-Modifiye push up test | up to 6 months
  The 30-second Modified Push-up Test measures core strength. The person starts in a push-up position but with knees on the floor. They perform as many push-ups as possible in 30 seconds, keeping the body straight and lowering the chest close to the ground. The score is the number of correct push-ups completed.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Kılınç, Principal Investigator — Hacettepe University; Özge Onursal Kılınç, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No